CLINICAL TRIAL: NCT06591429
Title: Investigation of Smoldering Inflammation in Multiple Sclerosis
Brief Title: Smoldering Inflammation in MS
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Matthew Brier, Assistant Professor of Neurology Adult, Neuroimmunology, Washington University School of Medicine
Other Study IDs: 202403168
Record Dates: First submitted 2024-09-07; First posted 2024-09-19 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Imaging; Inflammation
MeSH Terms: conditions — Multiple Sclerosis; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood and spinal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Adults with MS taking part in this study.
  Interventions: Radiation: Radiotracer [11C]-CS1P1; Radiation: Radiotracer [11C]-DPA-713; Drug: anti-CD20 MS treatment; Radiation: Radiotracer [12F]-FDG

INTERVENTIONS:
Radiation: Radiotracer [11C]-CS1P1 — Radiotracer used in PET/CT scans of the head and neck Dose range: 12-17 mCi
Radiation: Radiotracer [11C]-DPA-713 — Radiotracer used in PET/CT scans of the head and neck Dose range:15-20 mCi
Drug: anti-CD20 MS treatment — MS treatment taken indepenently after initial testing
Radiation: Radiotracer [12F]-FDG — used in PET/CT scans of the head and neck Dose: 5-7 mCi

SUMMARY:
The goal of this observational study is to learn about inflammation in those with relapsing remitting Multiple Sclerosis (MS). The main questions it aims to answer are:

* How does abnormal neural inflammation compare to cellular and molecular inflammation in MS?
* Once treated, why does abnormal inflammation persist?

DETAILED DESCRIPTION:
The purpose of this study is to combine multi-tracer PET and high-resolution CSF analysis to understand the inflammatory landscape of MS and to identify components of inflammation which do not resolve with high-efficacy DMT and are hypothesized to drive disability accumulation via smoldering inflammation. Identification of components of the pathologic cascade which do not respond to extant therapies will motivate future, complementary therapies targeted at yet untreated MS pathology.

Current MS disease modifying therapies (DMT) focus on reducing the inflammatory or auto-immune component of the disease. Highly effective DMTs are incredibly effective at reducing this inflammation such that new lesions and clinical relapses are increasingly rare. However, despite these advances, most patients will experience clinical worsening independent of relapse activity. This eventually manifests as progressive MS and stubbornly resists therapy. One hypothesized driver of this clinical progression is smoldering inflammation. Smoldering inflammation is defined as ongoing inflammation sufficient to cause accumulating tissue injury but insufficient to cause clinical relapse. The nature of this smoldering inflammation is poorly understood. Emerging imaging biomarkers have identified smoldering inflammation, but those markers are not well-linked to cellular mechanisms. A key innovation of this approach is that, by comparing pre- vs. post-treatment single-cell RNA sequencing data, the researchers will identify cell populations that are most sensitive and resistant to treatment and relate these findings to imaging changes. Identifying components of persistent inflammation may identify future treatment targets.

25 adult patients with relapsing remitting multiple sclerosis will be enrolled in this study. Patients will be recruited from the John L. Trotter MS Center at Washington University in St. Louis. Participants will be referred to the study by their treating neurologist.

[11C]-CS1P1 and [11C]-DPA-713 are the investigational radiotracers used in this study. Participation in this study consists of several visits. Visits include 1) (pre-)screening and clinical, 2) baseline lumbar puncture, 3) baseline [11C]-DPA-713 PET/CT, 4) baseline [11C]-CS1P1 PET/CT, 5) baseline [18F]-FDG PET/MRI, 6) follow-up lumbar puncture, 7) follow-up [11C]-DPA-713 PET/CT, 8) follow-up [11C]-CS1P1 PET/CT, and 9) follow-up [18F]-FDG PET/MRI. Baseline and follow-up visits of the same type (e.g., steps 3 and 7) are identical with baseline occurring at enrollment and follow-up occurring at least nine months but no more than 12 months after DMT initiation. Screening session must precede the clinical sessions. At each the baseline and follow-up time point, the lumbar puncture and each imaging session may occur in any order. At baseline and follow up, all sessions will take place within approximately 1 month. Multiple sessions can occur on the same day. Consecutive imaging sessions will be separated by 6 half-lives of the initially injected radiotracer.

This pilot study will link the molecular specificity and high spatial resolution of combined positron emission tomography and magnetic resonance imaging with the molecular explanatory power of single-cell RNA sequencing to investigate the effects of B cell depletion, or other similarly efficacious treatments, on smoldering inflammation and characterize the nature of persistent inflammation which contributes to disability in patients with MS. A key innovation of this approach is that, by comparing pre- vs. post-treatment single-cell RNA sequencing data, researchers will identify cell populations that are most sensitive and resistant to treatment and relate these findings to imaging changes. Identifying components of persistent inflammation may identify future treatment targets.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, any race
* Age ≥ 18 years
* Capable of providing written informed consent for volunteering to undergo research procedures
* Diagnosis of MS as established by the referring physician and confirmed by the Sponsor-Investigator. Only patients with active disease, defined as at least 1 enhancing lesion present in the preceding 6 months, will be enrolled
* Treatment naïve except for relapse-related treatments such as corticosteroids or plasmapheresis,
* Planned initiation, at the discretion of the referring physician, of a high efficacy DMT. High efficacy DMT will be defined to include ocrelizumab, natalizumab, or any MS treatment in the opinion of the Sponsor-Investigator to have similar efficacy as the named treatments
* Clinical labs, including at least a CBC and BMP, without significant abnormality as determined by the Sponsor-Investigator or designee, within the 3 months prior to enrollment

Exclusion Criteria:

* Presence of a low binding polymorphism for TSPO
* Hypersensitivity to [11C]-CS1P1, [11C]-DPA-713, [18F]-FDG, or any of their excipients
* Contraindications to PET, CT or MRI (e.g. certain incompatible electronic medical devices, inability to lie still for extended periods) that make it potentially unsafe for the individual to participate
* eGFR less than 60 (for gadolinium)
* Severe claustrophobia
* Women who are currently pregnant or breast-feeding
* Currently undergoing radiation therapy
* Insulin dependent diabetes
* Contraindication to lumbar puncture (LP), including use of antiplatelet therapy (other than aspirin 81mg), therapeutic anticoagulation, or space occupying intracranial mass. History of a coagulopathy is also exclusionary
* Any condition that, in the opinion of the Sponsor-Investigator or designee could increase risk to the participant, limit the participant's ability to tolerate the research procedures or interfere with collection of the data (e.g., renal or liver failure, advanced cancer)
* Current or recent (within 12 months prior to screening) participation in research studies involving radioactive agents such that the total research-related radiation dose to the participant in any given year would exceed 5 rem

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 25 adult patients with relapsing remitting multiple sclerosis will be enrolled in this study. Patients will be recruited from the John L. Trotter MS Center at Washington University in St. Louis. Participants will be referred to the study by their treating neurologist.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Volume of Distribution (Vt) of DPA-713 and CS1P1 and Cerebral metabolic rate of glucose (CMRglc) in white matter lesions and normal appearing white matter before and after treatment. | 1 year
Changes in scRNAseq measures of inflammatory cell types in the CSF before and after treatment | 1 year

SECONDARY OUTCOMES:
Correlation between changes in Vt or CMRglc compared to changes in cell type numbers from scRNAseq | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Barnes Jewish Center for Clinical Imaging Research, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Hauser SL, Bar-Or A, Comi G, Giovannoni G, Hartung HP, Hemmer B, Lublin F, Montalban X, Rammohan KW, Selmaj K, Traboulsee A, Wolinsky JS, Arnold DL, Klingelschmitt G, Masterman D, Fontoura P, Belachew S, Chin P, Mairon N, Garren H, Kappos L; OPERA I and OPERA II Clinical Investigators. Ocrelizumab versus Interferon Beta-1a in Relapsing Multiple Sclerosis. N Engl J Med. 2017 Jan 19;376(3):221-234. doi: 10.1056/NEJMoa1601277. Epub 2016 Dec 21. PMID 28002679
- [Result] Maggi P, Sati P, Nair G, Cortese ICM, Jacobson S, Smith BR, Nath A, Ohayon J, van Pesch V, Perrotta G, Pot C, Theaudin M, Martinelli V, Scotti R, Wu T, Du Pasquier R, Calabresi PA, Filippi M, Reich DS, Absinta M. Paramagnetic Rim Lesions are Specific to Multiple Sclerosis: An International Multicenter 3T MRI Study. Ann Neurol. 2020 Nov;88(5):1034-1042. doi: 10.1002/ana.25877. Epub 2020 Sep 9. PMID 32799417
- [Result] Endres CJ, Pomper MG, James M, Uzuner O, Hammoud DA, Watkins CC, Reynolds A, Hilton J, Dannals RF, Kassiou M. Initial evaluation of 11C-DPA-713, a novel TSPO PET ligand, in humans. J Nucl Med. 2009 Aug;50(8):1276-82. doi: 10.2967/jnumed.109.062265. Epub 2009 Jul 17. PMID 19617321
- [Result] Brier MR, Hamdi M, Rajamanikam J, Zhao H, Mansor S, Jones LA, Rahmani F, Jindal S, Koudelis D, Perlmutter JS, Wong DF, Nickels M, Ippolito JE, Gropler RJ, Schindler TH, Laforest R, Tu Z, Benzinger TLS. Phase 1 Evaluation of 11C-CS1P1 to Assess Safety and Dosimetry in Human Participants. J Nucl Med. 2022 Nov;63(11):1775-1782. doi: 10.2967/jnumed.121.263189. Epub 2022 Mar 24. PMID 35332093
- [Result] Lassmann H, van Horssen J, Mahad D. Progressive multiple sclerosis: pathology and pathogenesis. Nat Rev Neurol. 2012 Nov 5;8(11):647-56. doi: 10.1038/nrneurol.2012.168. Epub 2012 Sep 25. PMID 23007702
- [Result] Hemond CC, Baek J, Ionete C, Reich DS. Paramagnetic rim lesions are associated with pathogenic CSF profiles and worse clinical status in multiple sclerosis: A retrospective cross-sectional study. Mult Scler. 2022 Nov;28(13):2046-2056. doi: 10.1177/13524585221102921. Epub 2022 Jun 24. PMID 35748669
- [Result] Mahad DH, Trapp BD, Lassmann H. Pathological mechanisms in progressive multiple sclerosis. Lancet Neurol. 2015 Feb;14(2):183-93. doi: 10.1016/S1474-4422(14)70256-X. PMID 25772897